CLINICAL TRIAL: NCT05830201
Title: The Presence of a Therapy Dog Reduces Pain and Anxiety During Pediatric Elbow Pin Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael J. Conklin, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300010224; UAB (Other: UAB)
Record Dates: First submitted 2023-03-03; First posted 2023-04-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Elbow Injury
MeSH Terms: conditions — Elbow Injuries

STUDY DESIGN:
Intervention Model Description: control group or therapy group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Dog will not be in room when child has elbow pins removed
  Interventions: Behavioral: No Dog Present
- Therapy Dog Group (Experimental): The dog will come in a few minutes before to meet with you and your child and ensure ease. The therapy dog will be present throughout the procedure and is able to sit on the exam table if desired.
  Interventions: Behavioral: Dog is Present

INTERVENTIONS:
Behavioral: No Dog Present — Dog is not present during pin removal
  Arms: Control Group
Behavioral: Dog is Present — Dog is present during pin removal
  Arms: Therapy Dog Group

SUMMARY:
The purpose of this research study is to assess whether the presence of therapy dogs can reduce pain and anxiety in children ages 3 to 10 having pins removed from their elbow.

DETAILED DESCRIPTION:
This procedure is done in an outpatient clinic 3-4 weeks after the pins are placed and can be uncomfortable and cause anxiety in some patients. Therapy dogs are trained to sit calmly with a patient on or near the exam table as a distraction from procedures.

ELIGIBILITY:
Inclusion Criteria:

* presenting to clinic for elbow pin removal post elbow fracture surgery

Exclusion Criteria:

* dog allergy
* fear of dogs

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Response | 1 year
  Wong-Baker FACES scale, a validated scale for assessing pain in pediatric patients, will be used to compare pain response; The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst."

SECONDARY OUTCOMES:
Anxiety Response | 1 year
  anxiety response will be assessed with the Faces, Legs, Activity, Cry and Consolability (FLACC) Scale, This scale ranges from: 0 = Relaxed and comfortable ; 1-3 = Mild discomfort ; 4-6 = Moderate pain ; 7-10 = Severe discomfort/pain
Anxiety Response | 1 year
  anxiety response will be assessed with heart rate in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Michael Conklin, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No